CLINICAL TRIAL: NCT00003776
Title: A Phase II Window Study of Trimetrexate With Simultaneous Leucovorin Protection in the Treatment of Newly Diagnosed Patients With Metastatic Osteosarcoma
Brief Title: Combination Chemotherapy and Surgery in Treating Patients With Newly Diagnosed Metastatic Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-102; CDR0000066905 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1507
Record Dates: First submitted 1999-11-01; First posted 2004-08-18 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoma
Keywords: metastatic osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Filgrastim; Cisplatin; Doxorubicin; Ifosfamide; Leucovorin; Methotrexate; trimetrexate glucuronate; Surgical Procedures, Operative

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: leucovorin calcium
Drug: methotrexate
Drug: trimetrexate glucuronate
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug or combining chemotherapy with surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and surgery in treating patients who have newly diagnosed metastatic osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of oral trimetrexate glucuronate with simultaneous leucovorin calcium protection in patients with newly diagnosed metastatic osteogenic sarcoma. II. Evaluate the toxicity of this regimen when administered prior to and following standard chemotherapy in patients with osteogenic sarcoma. III. Correlate response with in vitro determinants of chemotherapy resistance in tumor samples obtained from these patients.

OUTLINE: Patients receive induction therapy of oral trimetrexate glucuronate (TMTX) and leucovorin calcium every 12 hours for 21 days (weeks 0-2). Patients receive leucovorin calcium for 3 additional days after the last dose of TMTX. If age prevents compliance with oral administration, patients receive TMTX IV and leucovorin calcium IV. Patients undergo definitive surgery 7-10 days after the induction therapy (week 4). Patients undergo surgery for metastatic disease, if indicated, as soon as possible following recovery from definitive surgery. Patients then receive maintenance therapy every 3 weeks for 8-9 months according to the following schedule: Patients receive ifosfamide IV over 1 hour 4 times daily on days 1-4 plus doxorubicin IV over 48 hours on days 1-2 in weeks 6, 14, and 22, and ifosfamide alone in week 30. Patients receive cisplatin IV over 4 hours for 1 day, plus doxorubicin IV over 48 hours for 2 days beginning on the same day as the first dose of cisplatin, in weeks 10, 18, and 26. Patients receive cisplatin alone in week 34. Patients receive filgrastim subcutaneously daily for 2 weeks starting 24 hours after the completion of each course of ifosfamide and cisplatin therapy. Patients receive methotrexate IV over 4 hours for 1 day, plus oral leucovorin calcium every 6 hours for at least 10 doses beginning 20 hours after the last dose of methotrexate, in weeks 9, 13, 17, 21, 25, 29, 33, and 37. In severe cases, patients receive leucovorin calcium IV over 24 hours. Patients who respond to induction therapy receive a second course of the same therapy in weeks 38-40. Patients are followed every 4 months for 1 year, then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 18-33 patients will be accrued for this study over 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, newly diagnosed (within one month of biopsy) malignant high grade osteosarcoma Must have pulmonary metastases (two or more nodules) and/or disease involving other bones or organs Must be an intent to resect at least one primary and/or metastatic site following preoperative chemotherapy Must have at least 1 evaluable site of disease No radiation induced sarcoma No osteosarcoma arising in premalignant bony lesions (e.g. Paget's disease)

PATIENT CHARACTERISTICS: Age: 30 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 3.0 times normal SGOT and/or SGPT less than 3.0 times normal Renal: Creatinine no greater than 1.5 times normal OR Creatinine clearance or radioisotope GFR greater than 70 mL/min Cardiovascular: Shortening fraction greater than 28% by echocardiogram OR Ejection fraction greater than 50% by radionuclide angiogram No history of pericarditis or myocarditis

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunomodulating agents except steroids Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: No concurrent immunomodulating agents except steroids Radiotherapy: No prior or concurrent radiotherapy Surgery: Prior biopsy only of primary or metastatic area No prior resection Other: No prior therapy for any other malignancy No concurrent co-trimoxazole

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-12; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gorlick, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States